CLINICAL TRIAL: NCT03823443
Title: COPD Exacerbation Blood and Urine Biomarkers Study
Status: Terminated | Type: Observational
Why Stopped: Difficulty enrolling
Sponsor: Columbia University (Other)
Collaborators: Alpha-1 Foundation (Other)
Responsible Party: Principal Investigator, Monica Goldklang, Assistant Professor of Medicine (in Anesthesiology), Columbia University
Other Study IDs: AAAR3691
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Acute Exacerbation Copd; Alpha-1 Anti-trypsin Deficiency
Keywords: exacerbation; cough; sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; alpha 1-Antitrypsin Deficiency; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and nasal swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This will be a prospective study examining serum levels of MMP-13 and alpha-1 antitrypsin as well as other biomarkers as well as urine biomarkers of smoking status and collagen degradation in the COPD patient population. Serum and urine biomarkers at baseline and after COPD exacerbations will be assessed against change in lung function as measured by pulmonary function testing.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD), a term describing emphysema and chronic bronchitis, is the third leading cause of death in the United States, with approximately 24 million US adults estimated to have the disease and over 130,000 US adults dying each year due to COPD. Acute exacerbations of chronic obstructive pulmonary disease (AECOPD), primarily the result of viral respiratory infections, result in accelerated decline in lung function and increased mortality. Recent work in our laboratory demonstrates that matrix metalloproteinase-13 (MMP-13), which has both collagenolytic and elastolytic activity, is increased in the bronchoalveolar lavage fluid of patients with COPD. It is well accepted that viral infections have significant consequences in smokers, particularly in patients with AATD related COPD.

COPD exacerbations clinically manifest with increased dyspnea, cough and sputum production, and from a societal cost standpoint are associated with significant increases in health care utilization. Recent data suggest that viral infections such as RSV increase MMP-13 secretion and expression within lung tissues. Therefore, the studies presented here seek to understand the effect of MMP-13 on COPD progression and the effect of disease exacerbations on MMP-13 and alpha-1 antitrypsin serum levels and later lung function decline. The investigators hypothesize that patients with COPD, in particular patients who fall into the "frequent exacerbator" phenotype (two or more exacerbations within the last year), will have increased levels of MMP-13 as compared to the general non-COPD patient population and that in the setting of a COPD exacerbation, levels will be increased. The investigators will assess how exacerbation MMP-13 levels predict later lung function decline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD (FEV1 <80% AND FEV1/FVC < 70%)
* Ages 35-80yrs

Exclusion Criteria:

* History of Asthma
* Bronchiectasis
* Carcinoma of the bronchus
* Recent COPD exacerbation or pulmonary infection (less than 1 month)
* Other significant respiratory disease
* Pregnancy

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population for this study will have a known diagnosis of COPD, confirmed by pulmonary function testing.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
MMP13 to Alpha-1 antitrypsin ratios | 1 year
  Serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Monica Goldklang, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States